CLINICAL TRIAL: NCT03709212
Title: Cultural Influences on Physical Activity and Exercise Beliefs in Patients With Chronic Kidney Disease
Acronym: CULTURE-CKD
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Kidney Care UK (Other); British Renal Society (Other)
Responsible Party: Sponsor
Other Study IDs: KCH-CULTURE CKD; 241792 (Other: IRAS number); KCH18-053 (Other: Sponsor site reference number (King's College Hospital))
Record Dates: First submitted 2018-08-08; First posted 2018-10-17 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Diseases; Physical Activity; Exercise Therapy
Keywords: Chronic Kidney Disease; Physical Activity; Cultural influences; Exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Individual semi-structured interview: 20 participants will undergo individual semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Participants will be recruited from three ethnic backgrounds; Black African/ Caribbean, South Asian and White Caucasian.
  Interventions: Other: interviews
- Focus Group 1: 10 participants female black African/ African Caribbean ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews
- Focus Group 2: 10 participants male Black African/ African Caribbean ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews
- Focus Group 3: 10 participants female South Asian ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews
- Focus Group 4: 10 participants male black South Asian ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews
- Focus Group 5: 10 participants female White Caucasian ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews
- Focus Group 6: 10 participants male White Caucasian ethnicity will undergo group semi-structured interviews to explore perceptions of living with Chronic Kidney Disease, attitudes and understanding of exercise and physical activity and any cultural influences that may influence attitudes or decisions regarding this.
  Interventions: Other: interviews

INTERVENTIONS:
Other: interviews — 20 participants will undergo individual semi-structured interviews, 60 will undergo one of 6 focus groups comprising of 10 participants of the same gender and ethnicity.
  Other Names: individual semi-structured; Focus groups

SUMMARY:
Cardiovascular disease (CVD) remains the leading cause of death in patients with Chronic Kidney Disease (CKD). Patients who spend a lot of time being inactive have an increased chance of developing CVD. Thus, interventions that can help to increase the levels of physical activity in patients with CKD are needed. A recent study the investigators completed with kidney transplant participants showed a benefit from the investigators supervised exercise programme. However, the investigators results showed that 11 of the 18 patients who dropped out from the 12-month study were from black and minority ethnic groups. Some patient feedback from these participants suggested that cultural beliefs; including women not being comfortable to exercise in front of men in an exercise class environment, and difficulties around appropriate dress for exercise classes, contributed to some of these participants' decisions to withdraw from the study. This has prompted the investigators to investigate, the cultural influences that may contribute to patient decisions about partaking in physical activity and exercise training. The aim of this study is therefore to invite patients with CKD from the three most widely represented ethnic groups found in our South-East London Hospital Trust (Black African and African-Caribbean; South Asian, and White Caucasian patients) to discuss their beliefs and the cultural influences that may affect their decision on whether to engage with exercise and physical activity. Participants will complete a questionnaire on physical activity levels, and a questionnaire that looks at a patient's readiness to be involved in physical activity, prior to attending interviews or group discussions. The questionnaires will be translated for use with non-English speaking participants and will be used to ensure we get views on physical activity from those participants who are active and not, and ready to be involved in physical activity, and not. A combination of individual interviews and group discussions will then be used to explore the understanding of the terms 'physical activity' and 'exercise', and cultural barriers to participation. The investigators will have interpreters present for all discussions, undertaken in the community. The work from this pilot study will be used to inform and design a larger multi-centre study with an aim to design physical interventions that are culturally sensitive, and appropriate for all patients with CKD in the United Kingdom.

DETAILED DESCRIPTION:
Background:

This present study will utilise Stokol's Social Ecological Theory of Health Behaviour as the main theoretical framework. This multi-level Ecological theory suggests that an individual's behaviour results from a complex interaction between the individual, the environment, and community in which they live. Multi-level theories are thought to be more robust and explanatory, in comparison to single-level approaches as they are representative of the public health approach to population change. Ecological approaches such as Stokol's Social Ecological Theory form a robust base to evaluate complex multifactorial behaviours such as physical activity. This theory has been used, and is promoted for use, in designing community-level health programmes, such as physical activity interventions for different ethnic communities. David Howe, a sports anthropologist, will advise the research team with the interpretation of the data using this framework.

Purpose:

The purpose of this present study is to utilise a mixed-methods design to explore the understanding of physical activity and exercise, and factors that contribute to a decision to be physically active or sedentary, in patients with CKD from different ethnic backgrounds. The investigators intend to measure self-reported physical activity levels with the General Practice Physical Activity Questionnaire (GPPAQ) and self-efficacy for exercise (readiness to start doing exercise) with Bandura's self-efficacy for exercise scale. The investigators then aim to explore perceptions, attitudes and values about physical activity and exercise therapy in different ethnic groups. The investigators will ensure that views are captured from patients stratified by activity, readiness to be active, age and gender. To accomplish these goals, the present study will explore: (i) the understanding of the terms 'physical activity' and 'exercise'; (ii) the interpretation of the socio-cultural contexts in which they choose (or not) to be physically active, and; (iii) the participants understanding of physical activity and exercise opportunities and barriers in their local environment. All questionnaires will be translated for non-English speaking participants, and individual and focus group discussions will be facilitated with translators.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of CKD that are representative of one of the 3 ethnic groups that will be studied (Black African and African-Caribbean; South Asian, and White Caucasian patients)
* Age > 18 years of age
* able to provide Informed consent

Exclusion Criteria:

* Uncontrolled medical condition (e.g. uncontrolled angina)
* Unstable psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to recruit up to 20 patients (for the individual interviews) and 60 patients (for the 6 single-sex focus groups), aged over 18 years or over with CKD from the 3 identified ethnic groups, will be recruited to the study. Each patient must have met the inclusion and exclusion criteria at entry level to the study. For focus groups the investigators will aim to meet with six to twelve participants per group. Appropriate topic guides will be developed and discussed with the patient advisory group, and the steering group. The investigators will continue with individual interviews and focus groups until data saturation is reached, there is no new data, no new themes, no new coding and the investigators are able to replicate the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
One-to-one semi-structured interview to explore participants experiences of living with Chronic Kidney Disease. | Through study completion, an average of one year
  To establish challenges and perceptions of living with this long term condition and how this has an impact on day to day life.
One-to-one semi-structured interview to explore participants experience of exercise and physical activity | Through study completion, an average of one year
  Any difficulties/ barriers to exercise or physical activity determined by a qualitative interview.
  Experiences of the exercise and physical activity by a qualitative interview. Benefits to under taking physical activity and exercise by a qualitative interview.
  Facilities and opportunities available to undertake exercise of physical activity by a qualitative interview.
  Any cultural influences that may have influenced decisions to participate in physical activity and exercise by a qualitative interview.

SECONDARY OUTCOMES:
Physical activity through General Practice Physical Activity Questionnaire (GPPAQ) | Through study completion, an average of one year
  GPPAQ is a reliable and validated questionnaire used to measure adult physical activity levels.
  It contains seven questions and provides a simple, 4-level Physical Activity Index (PAI) of: Active, Moderately Active, Moderately Inactive, and Inactive.
  PAI scale from question answers range from 'inactive' which indicates a sedentary job and no physical exercise or cycling. This scale then ranges through to 'active' indicates a sedentary job and ≥ 3 hours physical exercise OR a standing job and 1-2.9 hours physical exercise per week OR a physical job and some but < 1 hour physical exercise per week.
  The classification of Physical Activity Index gives an indication of how active an adult individual is on a weekly basis.
Self-efficacy to regulate exercise | Through study completion, an average of one year
  Bandura self-efficacy for exercise scale
  This questionnaire contains 18 questions to answer with regards to self-efficacy to exercise on a scale of 0-100.
  The questions relate to the certainty of the participant to continue with a regular exercise routine (three or more times a week) in relation to the questions posed.
  In relation to the scale 0 is 'cannot do at all' and 100 is 'highly certain can do'.
  The total score is calculated by summing the responses to each question. The scale has a range of total scores from 0-1,800. A higher score indicates greater exercise related self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene A Greenwood, PhD, BSc, Study Chair — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study group plans to make anonymised data available as supplementary text when the study is published as an online manuscript. For example Plos one
Supporting Information: Study Protocol, SAP
Time Frame: within 12 months of study completion
Access Criteria: with open access publication

REFERENCES:
- [Derived] Mayes J, Castle EM, Greenwood J, Ormandy P, Howe PD, Greenwood SA. Cultural influences on physical activity and exercise beliefs in patients with chronic kidney disease: 'The Culture-CKD Study'-a qualitative study. BMJ Open. 2022 Jan 11;12(1):e046950. doi: 10.1136/bmjopen-2020-046950. PMID 35017229